CLINICAL TRIAL: NCT06806124
Title: Analysis of Hematological Biomarkers, Muscle Respiratory Function and Sports Performance in CrossFit® Athletes Using the Elevation Training Mask 2.0 Upon Return to a High-intensity Training Program After Recovering from COVID-19. a Single-blind, Multicenter, Randomized Clinical Trial.
Brief Title: Impact of the Elevation Training Mask in CrossFit® Post-SARS-CoV-2 Infection.
Acronym: ETMEXCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Diego Fernández Lázaro, Professor and Researcher, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI 19-1361
Record Dates: First submitted 2025-01-25; First posted 2025-02-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: COVID19- Infection with SARS-CoV-2 Virus; SARS-CoV-2 Positive Patients; COVID-19 Pulmonary Complications; SARS-CoV-2 Infection (Symptomatic)
Keywords: Elevation Training Mask; SARS-CoV-2; CrossFit®; Spirometric Parameters; Hematological Biomarkers; WOD
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The first week, the additional altitude simulation was 914 m and in the second, 1,829 m. These initial 2 weeks served to adjust the use of the The Elevation Training Mask (ETM) 2.0 during training, as a process of acclimatization to the altitude simulation and airflow restriction. For the period between weeks 3 and 6 (both inclusive) the simulated altitude was 2,743 m, and for weeks 7-12 (both inclusive), the ETM was set to simulate 3658 m altitude
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elevation Training Mask (ETM) Group (Experimental): Elevation Training Mask (ETM) using the corresponding air restriction openings and filters. The first week, the additional altitude simulation was 914 m and the second, 1,829 m. These initial 2 weeks served to familiarize to the use of the ETM during training, as a process of acclimatization to the altitude simulation and airflow restriction. For the period between weeks 3 and 6 (both included) the simulated altitude was 2,743 m, and for weeks 7-12 (both included), the ETM was set to simulate 3,658 m altitude.
  Interventions: Device: Elevation Training Mask
- Control Group (Sham Comparator): For the Control Group, the Elevation Training Mask (ETM) was used for 12 weeks with the largest openings available and without using the air restriction filters, so that there was little respiratory obstruction but the reduction in air flow was minimal, with the aim of having a simulated ETM treatment.
  Interventions: Device: Sham Elevation Training Mask

INTERVENTIONS:
Device: Elevation Training Mask — The Elevation Training Mask (ETM) 2.0 was used in all 36 training sessions over the 12 weeks of the study with progressive increases in air restriction to simulate altitude training. This methodology of using ETM during exercise was chosen following the study by Porcari et al. The first week, the additional altitude simulation was 914 m and in the second, 1,829 m. These initial 2 weeks served to adjust the use of the ETM during training, as a process of acclimatization to the altitude simulation and airflow restriction. For the period between weeks 3 and 6 (both inclusive) the simulated altitude was 2,743 m, and for weeks 7-12 (both inclusive), the ETM was set to simulate 3658 m altitude.
  Other Names: Experimental Group
  Arms: Elevation Training Mask (ETM) Group
Device: Sham Elevation Training Mask — For the Control Group, the Elevation Training Mask (ETM) 2.0 was used for 12 weeks with the largest openings available and without using the air restriction filters, so that there was little respiratory obstruction and the reduction in air flow was minimal, with the aim of having a simulated ETM treatment
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
Introduction: The Elevation Training Mask (ETM) could restore respiratory or hematological organic damages from the acute or post-infection phase of severe acute respiratory syndrome coronavirus 2 (SARSCoV2) because it would allow the application of hypoxia and respiratory muscle training during exercise. The aim of this study was to comparatively evaluate the respiratory and hematological parameters and performance of athletes who resume CrossFit® training using the ETM with respect to a control group (CG).

Material and methods: A single-blind randomized clinical trial, following the CONSORT ("Consolidated Standards of Reporting Trials") recommendations, 20 trained male athletes were randomly assigned to an experimental group (EG) using the ETM and to a CG using the simulated ETM, they completed 12 weeks of CrossFit® training after 1 month of the cessation of SARS-CoV-2 symptoms. Pre- and post-training tests included spirometric, hematological, and sports performance assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 to 50 years.
* Autonomy in training activities of CrossFit® programs, at least 1 month after the cessation of symptoms of SARS-CoV-2 infection -2 infection.
* No hospitalization for COVID-19.
* Autonomy in training activities of CrossFit® programs, at least 1 month after the cessation of symptoms of SARS-CoV-2 infection, to avoid residual effects of the disease and increase the safety of the athlete.
* ≥20 months of experience training CrossFit®.
* ≥2 participations in CrossFit® competitions in the last season.
* Having completed Fran WODs ≤ 250 seconds before suffering from COVID-19. - Passing a complete pre-study medical examination to rule out pre-existing diseases or injuries, insisting particularly on the cardio-pulmonary examination.-- No consumption of illegal drugs according to the World Anti-Doping Agency (WADA) (stimulants, blood derivatives, anabolic) or take drugs (e.g. tramadol) or other ergogenic products.
* Be informed about all possible risks or discomforts and benefits associated with the study and sign the informed consent form;.
* Health sports insurance coverage.

Exclusion Criteria:

* Included any renal dysfunction, recent febrile illness, lower limb trauma or any history of muscle injury.
* SARS-CoV-2 reinfection during the study.
* Recent exposure to an altitude stimulus or hypoxia, except for the altitude of their usual residence (1063 m in Soria and 798 m in Salamanca).
* Participants were also prevented to perform any intense physical activity outside the designed training protocol throughout the study and encouraged to follow the dietary instructions provided.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — volunteer male CrossFit® athletes
Enrollment: 20 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
maximum inspiratory pressure (MIP) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Maximal inspiratory pressure (MIP) evaluation in centimeters of water (cmH2O). MIP is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength.
maximum expiratory pressure (MEP) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Evaluation maximal expiratory pressure (MEP) aluation in centimeters of water (cmH2O). MEP measures the maximum positive pressure that can be generated from one expiratory effort starting from total lung capacity

SECONDARY OUTCOMES:
forced vital capacity (FVC) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Evaluation of Forced vital capacity (FVC) in Liters (L). FVC is a pulmonary function measurement that represents the total amount of air a person can forcibly exhale from their lungs after taking the deepest breath possible.
forced expiratory capacity in 1 second (FEV1) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Evaluation of forced expiratory capacity in 1 second (FEV1) in Liters (L). FEV1 indicates the volume of air a person can forcefully exhale in one second.
maximum voluntary ventilation (MVV) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Evaluation of Maximal Voluntary Ventilation (MVV) in Liters / minute (L/min). MVV is a measure of the maximum amount of air a person can breathe in and out within a specific time frame, typically one minute
vital capacity (VC) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Evaluation of vital capacity (VC) in in Liters (L).
red blood cells (RBC) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Erythrocytes, red blood cells (RBC), are the functional components of blood responsible for transporting gases and nutrients throughout the human body. Evaluation of RBC million / microliter (mill/µL).
Hemoglobin (Hb) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Hemoglobin (Hb) is the protein molecule in red blood cells that carries oxygen from the lungs to the body's tissues and returns carbon dioxide from the tissues back to the lungs. Hgb is made up of four protein molecules (globulin chains) that are connected. Evaluation of Hb in grams / deciliter (g/dL).
hematocrit (Hct) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  A hematocrit test (Hct) is a simple blood test that measures the percentage of red blood cells in your blood. Evaluation of Hct in Percentage (%).
reticulocytes (RET) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Reticulocytes are immature red blood cells (RBCs) produced in the bone marrow and released into the peripheral blood, where they mature into RBCs within 1 to 2 days. Evaluation of Reticulocytes in Percentage (%).
erythropoietin (EPO) | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Erythropoietin (EPO) is a hormone that regulates the production of red blood cells. It is produced by kidney cells in response to low oxygen levels in the tissues. EPO promotes the formation of red blood cells by the bone marrow. EPO deficiency can result in reduced production of red blood cells, leading to anemia. EPO is also known as eritropoyetina or hemopoyetina. Evaluation of EPO in milliunits/milliliter (mU/mL).

OTHER OUTCOMES:
Fran WOD | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Work of the Day (WOD): Perform the 21 Thrusters and 21 Pull-Ups, then 15 Thrusters and 15 Pull-Ups, then 9 Thrusters and 9 Pull-Ups, as fast as possible. Evaluation of Fran WOD in seconds (s).
CrossFit® Total | First day of study and after 12 weeks of Elevation Training Mask 2.0 use (end of study)]
  Work of the Day (WOD): Sum of the best of 3 attempts at each lift:
  Back Squat; Shoulder Press; Deadlift. Attempt each lift 3 times. The weight must increase after each successful attempt at each movement. The weight may not be decreased after the first attempt. A failed rep counts as an attempt. Take the Back Squat and Shoulder Press (aka: Strict Press) from the weight rack. Evaluation of CrossFit® Total in kilograms (Kg).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Fernández Lázaro, Vice Dean and Professor, Principal Investigator — Faculty of Health Sciences, University of Valladolid, Soria Campus (Spain)
Locations (1):
- Department of Cell Biology, Genetics, Histology and Pharmacology of the University of Valladolid, Soria, Soria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Lazaro D, Seco-Calvo J, Santamaria G, Donoso DJ, Roche E, Garrosa M. Twelve weeks of respiratory muscle training enhance respiratory function in CrossFit(R) athletes returning to exercise post-SARS-CoV-2 infection: single-blind randomized clinical trial. BMC Sports Sci Med Rehabil. 2025 Aug 14;17(1):236. doi: 10.1186/s13102-025-01261-9. PMID 40814059